CLINICAL TRIAL: NCT02766335
Title: A Phase II Study of MEDI4736 for Previously Treated Patients With Stage IV Squamous Cell Lung Cancer and No Matching Biomarkers (Lung-Map Sub-Study)
Brief Title: Lung-MAP: Durvalumab as Second-Line Therapy in Treating Patients With Recurrent Stage IV Squamous Cell Lung Cancer and No Matching Biomarkers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1400A; NCI-2014-01378 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1400A; S1400A (Other: SWOG); S1400A (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2016-05-06; First posted 2016-05-09 (Estimated); Results first posted 2021-12-30 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Recurrent Squamous Cell Lung Carcinoma; Stage IV Squamous Cell Lung Carcinoma AJCC v7
MeSH Terms: interventions — Docetaxel; durvalumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (MEDI4736 - closed to accrual 12/2015) (Experimental): Patients receive durvalumab IV over 60 minutes on day 1. Treatment repeats every 14 days for 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Other: Laboratory Biomarker Analysis
- Arm II (docetaxel - closed to accrual 4/2015) (Active Comparator): Patients receive docetaxel IV on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. (closed to accrual with Revision #2 4/22/15)
  Interventions: Drug: Docetaxel; Other: Laboratory Biomarker Analysis
- Arm III (MEDI4736 retreatment) (Experimental): For patients assigned to Arm 1, MEDI4736: Upon evidence of progression following discontinuation of 12 months of treatment, patients may restart treatment with Arm 3, MEDI4736 for up to 12 months with the same treatment guidelines followed during the initial 12-month treatment period. Patients will only be able to restart treatment once; thus a maximum of two 12-month periods will be allowed. Patients receive durvalumab IV over 60 minutes on day 1. Treatment repeats every 14 days for 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Arm II (docetaxel - closed to accrual 4/2015)
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
  Arms: Arm I (MEDI4736 - closed to accrual 12/2015); Arm III (MEDI4736 retreatment)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well durvalumab works in treating patients with stage IV squamous cell lung cancer that has come back after previous treatment. This is a "non-match" sub-study that includes all screened patients not eligible for a biomarker-driven sub-study. Monoclonal antibodies, such as durvalumab, may be able to shrink tumors. Durvalumab may be effective in treating patients with squamous cell lung cancer.

DETAILED DESCRIPTION:
CO-PRIMARY OBJECTIVES:

I. To assess the response rate (confirmed and unconfirmed, complete and partial) among patients treated with durvalumab (MEDI4736).

II. To assess the response rate (confirmed and unconfirmed, complete and partial) among programmed death ligand 1 (PD-L1) positive patients treated with MEDI4736.

SECONDARY AND EXPLORATORY OBJECTIVES:

I. To assess investigator-assessed progression-free survival (IA-PFS) among patients treated with MEDI4736.

II. To assess IA-PFS among PD-L1 positive patients treated with MEDI4736. III. To assess overall survival (OS) in patients treated with MEDI4736. IV. To assess overall survival (OS) in PD-L1 positive patients treated with MEDI4736.

V. To evaluate the frequency and severity of toxicities associated with MEDI4736.

VI. To assess immune-related IA-PFS using a modified response criteria adapted for immunotherapy (immune-related response criteria [irRC]-IA-PFS) in all patients and in the subset of patients determined to be PD-L1 positive treated with MEDI4736.

VII. To compare IA-PFS, irRC-IA-PFS, OS, toxicity and response rates between patients randomized to MEDI4736 versus docetaxel.

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To identify additional predictive or prognostic tumor/blood biomarkers beyond the chosen biomarker.

II. To identify potential resistance biomarkers at disease progression. III. To establish a tissue/blood repository from patients with refractory squamous cell cancer.

MEDI4736 RE-TREATMENT OBJECTIVES:

I. To evaluate response rates (confirmed and unconfirmed, complete and partial responses) among patients re-treated with MEDI4736.

II. To estimate median PFS from the date of re-treatment.

OUTLINE (CLOSED TO ACCRUAL 12/18/2015):

Patients with tumors that do not match one of the currently active drug-biomarker combinations receive durvalumab intravenously (IV) over 60 minutes on day 1. Courses repeat every 2 weeks for 12 months in the absence of disease progression or unacceptable toxicity. Upon evidence of progression following discontinuation of 12 months of treatment, patients may restart treatment and continue for up to 12 additional months (Arm III).

ARM I: (Closed to accrual 12/2015) Patients receive durvalumab intravenously (IV) over 60 minutes on day 1. Treatment repeats every 14 days for 12 months in the absence of disease progression or unacceptable toxicity.

ARM II (CLOSED TO ACCRUAL 4/2015): Patients receive docetaxel IV on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. (closed to accrual with Revision #2 4/22/15)

ARM III: For patients assigned to Arm 1, MEDI4736: Upon evidence of progression following discontinuation of 12 months of treatment, patients may restart treatment with Arm 3, MEDI4736 for up to 12 months with the same treatment guidelines followed during the initial 12-month treatment period. Patients will only be able to restart treatment once; thus a maximum of two 12-month periods will be allowed. Patients receive durvalumab IV over 60 minutes on day 1. Treatment repeats every 14 days for 12 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, all patients are followed up every 6 months for the first 2 years and then at the end of the year 3 from date of sub-study/re-registration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all SCREENING/PRE-SCREENING and SUB-STUDY REGISTRATION COMMON ELIGIBILITY CRITERIA as specified in S1400: Phase II/III Biomarker-Driven Master Protocol for Previously Treated Squamous Cell Lung Cancer (Lung-Map)
* Patients must have been assigned to S1400A
* Patients must not have any prior exposure to immunotherapy such as, but not limited to anti-programmed death 1 (PD-1) or anti-PD-L1 antibodies; prior exposure to the following is allowed: anti-cytotoxic T lymphocyte antigen 4 (CTLA-4) antibodies, live attenuated vaccines, anti-EGFR agents and sargramostim (GM-GSF)
* Patients must not have received nitrosoureas or mitomycin-C within 42 days prior to sub-study registration
* Patients must not have any active or prior documented autoimmune or inflammatory disease (including inflammatory bowel disease, diverticulitis with the exception of diverticulosis, celiac disease, irritable bowel disease; Wegener syndrome; Hashimoto syndrome) within 3 years prior to sub-study registration; patients with vitiligo, alopecia, Grave's disease, or psoriasis requiring systemic treatment within the past 3 years are not eligible
* Patients must not have any history of primary immunodeficiency
* Patients must not have received any immunosuppressive medication within 28 days prior to sub-study registration and must not be planning to receive any such agents while on protocol treatment; however, intranasal and inhaled corticosteroids or systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent are allowed
* Patients must not have any prior grade >= 3 immune-related adverse event (irAE) or any unresolved irAE > grade 1
* Patients must not have any history of organ transplant that requires use of immunosuppressives
* Patients must not have any known allergy or reaction to any component of the MEDI4736 formulation
* Patients must not have a known history of tuberculosis
* Patients must not have received a live attenuated vaccination within 28 days prior to sub-study registration
* Patients must not have known human immunodeficiency virus (HIV), hepatitis B or C positivity
* Patients must also be offered participation in banking for future use of specimens
* STEP 2 TO MEDI4736 RE-TREATMENT REGISTRATION:
* Patient must have progressed following 12 months of treatment with MEDI4736; patients who discontinue MEDI4736 prior to the completion of 12 months (for any reason) are not eligible; patients who have already completed two 12-month periods of treatment are not eligible
* Patients may have measurable or non-measurable disease documented by computed tomography (CT) or magnetic resonance imaging (MRI); the CT from a combined positron emission tomography (PET)/CT may be used to document only non-measurable disease unless it is of diagnostic quality; measurable disease must be assessed within 28 days prior to re-treatment registration; pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease; non-measurable disease must be assessed within 42 days prior to re-treatment registration; all disease must be assessed and documented on the Baseline Tumor Assessment Form; patients whose only measurable disease is within a previous radiation therapy port must demonstrate clearly progressive disease (in the opinion of the treating investigator) prior to RE-TREATMENT registration
* Patients must have a CT or MRI scan of the brain to evaluate for central nervous system (CNS) disease within 42 days prior to RE-TREATMENT registration; patient must not have leptomeningeal disease, spinal cord compression or brain metastases unless: metastases have been locally treated and have remained clinically controlled and asymptomatic for at least 14 days following treatment and prior to RE-TREATMENT registration, AND patient has no residual neurological dysfunction and has been off corticosteroids for at least 24 hours prior to RE-TREATMENT registration
* Patients must not have received any treatment after discontinuing MEDI4736 with the following exceptions; localized palliative radiation therapy is allowed for symptom management, provided and treatment is completed >= 14 days prior to RE-TREATMENT registration; local treatment for brain metastases is allowed
* Patients must not have received any immunosuppressive medication within 28 days prior to RE-TREATMENT registration and must not be planning to receive any such agents while on protocol treatment; however, intranasal and inhaled corticosteroids or systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent are allowed
* Patients must not have any prior grade >= 3 immune-related adverse event (irAE) or any unresolved irAE > grade 1 (MEDI4736 RE-TREATMENT)
* Patients must not have received a live attenuated vaccination within 28 days prior to RE-TREATMENT registration
* Patients must not have known HIV, hepatitis B or hepatitis C positivity
* Patients must not be planning to receive any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment; concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable
* Absolute neutrophil count (ANC) >= 1,500/mcl obtained within 28 days prior to RE-TREATMENT registration
* Platelet count >= 100,000 mcl obtained within 28 days prior to RE-TREATMENT registration
* Hemoglobin >= 9 g/dL obtained within 28 days prior to RE-TREATMENT registration
* Serum bilirubin =< institutional upper limit of normal (IULN) within 28 days prior to RE-TREATMENT registration; for patients with liver metastases, bilirubin must be =< 5 x IULN
* Either alanine aminotransferase (ALT) or aspartate aminotransferase (AST) =< 2 x IULN within 28 days prior to RE-TREATMENT registration (if both ALT and AST are done, both must be =< 2 IULN); for patients with liver metastases, either ALT or AST must be =< 5 x IULN (if both ALT and AST are done, both must be =< 5 x IULN)
* Patients must have a serum creatinine =< the IULN OR measured or calculated creatinine clearance >= 50 mL/min using the Cockcroft-Gault formula
* Patients must have Zubrod performance status of 0-1 documented within 28 days prior to RE-TREATMENT registration
* Prestudy history and physical exam must be obtained within 28 days prior to RE-TREATMENT registration
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* Patients with impaired decision-making capacity are eligible as long as their neurological or psychological condition does not preclude their safe participation in the study (e.g., tracking pill consumption and reporting adverse events to the investigator)
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2014-07-31 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vassiliki Papadimitrakopoulou, Principal Investigator — SWOG Cancer Research Network
Locations (993):
- United States (993):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Yuma Cancer Center, Yuma, Arizona
  - Mercy Cancer Center-Hot Springs, Hot Springs, Arkansas
  - Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Hospital, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente, Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Feather River Cancer Center, Paradise, California
  - PCR Oncology, Pismo Beach, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Northbay Cancer Center, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Memorial Hospital Central, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Medical Oncology and Hematology Group PC-Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale-New Haven Hospital Saint Raphael Campus, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Charlotte Hungerford Hospital Center for Cancer Care, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Low Country Cancer Care Associates PC, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Leeward, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Hines Veterans Administration Hospital, Hines, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Hematology Oncology Consultants Limited, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Michiana Hematology Oncology PC-Crown Point, Crown Point, Indiana
  - IU Health Central Indiana Cancer Centers-Fishers, Fishers, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Covenant Medical Center, Waterloo, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Newman Regional Health, Emporia, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Medical Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Hardin Memorial Hospital, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Norton Suburban Hospital and Medical Campus, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Medical Oncology LLC, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Mary Bird Cancer Center/Saint Tammany Parish, Covington, Louisiana
  - Mary Bird Perkins Cancer Center/Terrebonne General Medical Center, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - West Jefferson Medical Center, Marrero, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - Robert Veith MD LLC, Metairie, Louisiana
  - University Health-Conway, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - LSU Healthcare Network/Saint Charles, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Mercy Hospital, Portland, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Western Maryland Regional Medical Center, Cumberland, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Montgomery General Hospital-Olney, Olney, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Winchester Hospital, Winchester, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Veteran's Administration Medical Center - Ann Arbor, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Botsford General Hospital, Farmington, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Point, Grosse Pointe, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mid-Michigan Medical Center - Midland, Midland, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Assarian Cancer Center, Novi, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon and Rectal Association, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Hematology Oncology Consultants PC, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Providence Hospital-Southfield Cancer Center, Southfield, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Baptist Cancer Center-Golden Triangle, Columbus, Mississippi
  - Boston Baskin Cancer Center-Grenada, Grenada, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Family Cancer Center-Oxford, Oxford, Mississippi
  - Family Cancer Center-Southhaven, Southaven, Mississippi
  - Baptist Memorial Hospital-Desoto, Southhaven, Mississippi
  - Baptist Cancer Institute-Starkville, Starkville, Mississippi
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - CoxHealth Cancer Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-North, Kansas City, Missouri
  - The University of Kansas Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Faith Regional Medical Offices West, Norfolk, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hemotology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Oncology Hematology West, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center, Scottsbluff, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology - Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Specialists-Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - 21st Century Oncology - Vegas Tenaya, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Alpine Hematology-Oncology, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Reno Oncology Consultants, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Ocean Medical Center, Brick, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Southern Ocean County Medical Center, Manahawkin, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - New York Oncology Hematology PC -Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Beth Israel Medical Center, New York, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Asheville Hematology-Oncology Associates, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - Hayworth Cancer Center, High Point, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Lake Norman Hematology Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Specialists-Matthews, Matthews, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Lake Norman Hematology Oncology Specialists-Mooresville, Mooresville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OneHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Ireland Cancer Center Landerbrook Health Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center Ireland Cancer Center, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Ireland Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - University Pointe, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH-Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - PinnacleHealth Cancer Center-Community Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates-Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates PA-St. Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Georgetown Hospital System, Georgetown, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Boston Baskin Cancer Center-Bartlett, Bartlett, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - Family Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Texas Oncology at Baylor Charles A Sammons Cancer Center, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - The Methodist Hospital System, Houston, Texas
  - MD Anderson Regional Care Center-Katy, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - MD Anderson Regional Care Center-Bay Area, Nassau Bay, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson Regional Care Center-Sugar Land, Sugar Land, Texas
  - MD Anderson Regional Care Center-The Woodlands, The Woodlands, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Memorial Hospital Of Martinsville, Martinsville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology Associates PC, Winchester, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Seattle Cancer Care Alliance at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Spokane Valley Cancer Center-Mayfair, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston, Charleston, West Virginia
  - WVUH-East City Hospital, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology SC-Appleton, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - The Alyce and Elmore Kraemer Cancer Care Center, West Bend, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Saint Clare's Hospital, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Arm 1: 78 participants randomized to the durvalumab arm, 9 ineligible and 1 did not receive any treatment. Thus 68 were eligible and evaluable for analyses. 4 participants were re-registered after progression to receive additional treatment with MEDI4736
  Arm 2: 38 participants randomized to the docetaxel arm, 30 were eligible and evaluable for analyses due to 2 being ineligible and 6 not receiving any protocol treatment.
Groups:
- Arm I (MEDI4736 - Closed to Accrual 12/2015): Participants receive durvalumab IV over 60 minutes on day 1. Treatment repeats every 14 days for 12 months in the absence of disease progression or unacceptable toxicity.
  Durvalumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
- Arm II (Docetaxel - Closed to Accrual 4/2015): Participants receive docetaxel IV on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. (closed to accrual with Revision #2 4/22/15)
  Docetaxel: Given IV
  Laboratory Biomarker Analysis: Correlative studies
- Arm III - MEDI4736 Retreatment: For participants assigned to Arm 1, MEDI4736: Upon evidence of progression following discontinuation of 12 months of treatment, participants may restart treatment with Arm 3, MEDI4736 for up to 12 months with the same treatment guidelines followed during the initial 12-month treatment period. Participants will only be able to restart treatment once; thus a maximum of two 12-month periods will be allowed. Participants receive durvalumab IV over 60 minutes on day 1. Treatment repeats every 14 days for 12 months in the absence of disease progression or unacceptable toxicity.
  Durvalumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
Period: Initial Registration
Arm/Group | Arm I (MEDI4736 - Closed to Accrual 12/2015) | Arm II (Docetaxel - Closed to Accrual 4/2015) | Arm III - MEDI4736 Retreatment
Started | 68 | 30 | 0
Eligible Participants Enrolled Before Docetaxel Arm Closed | 32 | 30 | 0
Completed | 10 | 0 | 0
Not Completed | 58 | 30 | 0
Not completed — Adverse Event | 6 | 3 | 0
Not completed — Refusal unrelated to adverse event | 1 | 0 | 0
Not completed — Progression/relapse | 49 | 15 | 0
Not completed — Death | 1 | 3 | 0
Not completed — not protocol specified | 1 | 9 | 0
Period: Re-registration of Arm I to MEDI4738
Arm/Group | Arm I (MEDI4736 - Closed to Accrual 12/2015) | Arm II (Docetaxel - Closed to Accrual 4/2015) | Arm III - MEDI4736 Retreatment
Started | 0 | 0 | 4
Completed | 0 | 0 | 2
Not Completed | 0 | 0 | 2
Not completed — Death | 0 | 0 | 1
Not completed — Progression/relapse | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (MEDI4736 - Closed to Accrual 12/2015) | Arm II (Docetaxel - Closed to Accrual 4/2015) | Total
Number analyzed (Participants) | 68 | 30 | 98
Age, Continuous [Median (Full Range); unit: years] | 66 [35 to 92] | 71 [50 to 83] | 67.3 [35 to 92]
Age, Customized [Count of Participants; unit: Participants]
  >=65 years | 36 | 21 | 57
  <65 years | 32 | 9 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 10 | 37
  Male | 41 | 20 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race and ethnicity may overlap in some patients, so total sum of categories may be greater than total number of participants.
  Participants
    White | 55 | 27 | 82
    Black | 6 | 1 | 7
    Asian | 5 | 1 | 6
    Multi-racial | 0 | 1 | 1
    Unknown race | 2 | 0 | 2
    Hispanic | 2 | 0 | 2
Number of lines of prior therapy for stage IV disease [Count of Participants; unit: Participants] — Population: While the docetaxel arm was enrolling, the eligibility stated that patients must have received exactly 1 line of prior therapy for stage IV disease or platinum-based chemotherapy for stage I-III disease with progression within a year of completing therapy. Therefore, the number of lines of prior therapy for stage IV disease was not captured prior to the revision in May 2015 that closed the docetaxel arm to accrual.
  Participants
    number analyzed (Participants) | 68 | 0 | 68
    0 | 16 |  | 16
    1 | 39 |  | 39
    2 | 11 |  | 11
    3+ | 2 |  | 2
Zubrod performance status [Count of Participants; unit: Participants] — 0- fully active, able to carry out all pre-disease performance without restriction
  1. restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    0 | 18 | 10 | 28
    1 | 42 | 16 | 58
    2 | 8 | 4 | 12
Weight loss in past 6 months [Count of Participants; unit: Participants]
  <5% | 48 | 29 | 77
  5%-10% | 12 | 1 | 13
  10%-<20% | 6 | 0 | 6
  >=20% | 2 | 0 | 2
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 17 | 6 | 23
  Former smoker | 47 | 21 | 68
  Never smoker | 4 | 3 | 7
Brain metatases reported at baseline [Count of Participants; unit: Participants]
  Yes | 4 | 1 | 5
  No | 64 | 29 | 93
Programmed death-ligand 1 (PD-L1) [Count of Participants; unit: Participants] — PD-L1 testing was only performed on participants on the durvalumab arm who had evaluable tissue. Population: PD-L1 testing was done for 43 participants on the durvalumab arm who had evaluable tissue samples.
  PD-L1 testing was not performed for participants on the docetaxel arm.
  Participants
    number analyzed (Participants) | 43 | 0 | 43
    >= 25 (positive) | 14 |  | 14
    < 25 (negative) | 29 |  | 29

OUTCOME MEASURES:

1. Primary Outcome: Response Rate in MEDI4736-treated Participants
Description: The percentage of participants with confirmed and unconfirmed, partial response and complete response to treatment with MEDI4736 per Response Evaluation Criteria in Solid Tumors Criteria (RECIST 1.1).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 3 years post registration
Population: Eligible and evaluable participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm I (MEDI4736 - Closed to Accrual 12/2015): Participants receive MEDI4736 (durvalumab) IV over 60 minutes on day 1. Treatment repeats every 14 days for 12 months in the absence of disease progression or unacceptable toxicity.
  Durvalumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Arm I (MEDI4736 - Closed to Accrual 12/2015)
Number analyzed (Participants) | 68
percentage of participants | 16 [7 to 25]

2. Primary Outcome: Overall Response Rate Among PD-L1 Positive Participants Treated With MEDI4736
Description: The percentage of PD-L1 positive participants with confirmed and unconfirmed, partial response and complete response to treatment with MEDI4736 per Response Evaluation Criteria in Solid Tumors Criteria (RECIST 1.1).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 3 years post registration
Population: PD-L1 positive participants treated with MEDI4736
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (MEDI4736 - Closed to Accrual 12/2015)
Number analyzed (Participants) | 14
percentage of participants | 14 [0 to 33]

3. Secondary Outcome: Investigator-assessed Progression-free Survival in Participants Treated With MEDI4736
Description: Duration from date of sub-study registration to date of first documentation of progression, per RECIST 1.1, assessed by local review or symptomatic deterioration, or death due to any cause.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions or an absolute increase of >= 0.5cm, or a measurable increase in a non-target lesion, or the appearance of new lesions or death due to disease without prior documentation of progression or symptomatic deterioration.
Time Frame: Up to 3 years post registration
Population: Eligible and evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (MEDI4736 - Closed to Accrual 12/2015)
Number analyzed (Participants) | 68
months | 2.9 [2.0 to 4.0]

4. Secondary Outcome: Investigator-assessed Progression-free Survival in PD-L1 Positive Participants Treated With MEDI4736
Description: Duration from date of sub-study registration to date of first documentation of progression, per RECIST 1.1, assessed by local review or symptomatic deterioration or death due to any cause.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions or an absolute increase of >= 0.5cm, or a measurable increase in a non-target lesion, or the appearance of new lesions or death due to disease without prior documentation of progression or symptomatic deterioration.
Time Frame: up to 3 years post registration
Population: Eligible and evaluable PD-L1 positive participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (MEDI4736 - Closed to Accrual 12/2015)
Number analyzed (Participants) | 14
months | 2.3 [1.4 to 4.2]

5. Secondary Outcome: Overall Survival in MEDI4736-treated Participants
Description: Duration from date of sub-study registration (or date of screening/pre-screening registration if patient never enrolls in a sub-study) to date of death due to any cause.
Time Frame: Up to 3 years post-registration
Population: Eligible and evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (MEDI4736 - Closed to Accrual 12/2015)
Number analyzed (Participants) | 68
months | 11.6 [10.2 to 14.3]

6. Secondary Outcome: Overall Survival in PD-L1 Positive MEDI4736-treated Participants
Description: as for outcome 5
Time Frame: up to 3 years post registration
Population: Eligible and evaluable PD-L1 positive participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (MEDI4736 - Closed to Accrual 12/2015)
Number analyzed (Participants) | 14
months | 10.7 [9.2 to 14.3]

7. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 5.0 for serious adverse events only and CTCAE Version 4.0 for routine toxicity reporting. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Population: Participants who received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Arm/Group | Arm I (MEDI4736 - Closed to Accrual 12/2015) | Arm II (Docetaxel - Closed to Accrual 4/2015)
Number analyzed (Participants) | 68 | 30
Participants
  Abdominal pain | 1 | 0
  Alanine aminotransferase increased | 2 | 1
  Anemia | 4 | 5
  Aspartate aminotransferase increased | 2 | 0
  Bone pain | 1 | 0
  Bronchopulmonary hemorrhage | 1 | 0
  Dehydration | 0 | 1
  Diarrhea | 0 | 1
  Dyspnea | 6 | 2
  Ejection fraction decreased | 1 | 0
  Fatigue | 3 | 5
  Febrile neutropenia | 0 | 3
  Gastrointestinal disorders - Other, specify | 0 | 1
  Generalized muscle weakness | 0 | 1
  Hypercalcemia | 1 | 0
  Hyperglycemia | 0 | 1
  Hyponatremia | 3 | 1
  Hypoxia | 2 | 1
  Immune system disorders - Other, specify | 0 | 1
  Infusion related reaction | 1 | 0
  Leukocytosis | 1 | 0
  Lung infection | 1 | 2
  Lymphocyte count decreased | 3 | 7
  Mucositis oral | 0 | 1
  Nausea | 1 | 0
  Neutrophil count decreased | 0 | 10
  Pneumonitis | 0 | 1
  Resp, thoracic and mediastinal disorders - Other | 0 | 1
  Sepsis | 0 | 2
  Stevens-Johnson syndrome | 0 | 1
  Syncope | 1 | 0
  Thromboembolic event | 0 | 1
  Urinary tract infection | 1 | 0
  Weight loss | 1 | 0
  White blood cell decreased | 0 | 6

8. Secondary Outcome: Investigator-assessed Progression-free Survival Assessed Using a Modified Response Criteria Adapted for Immunotherapy in Participants Treated With MEDI4736
Description: Duration from date of sub-study registration to date of first documentation of immune related response criteria-progression assessed by local review or symptomatic deterioration (as defined above), or death due to any cause
Time Frame: up to 3 years post registration
Population: No data collected for this outcome measure
Arm/Group | Arm I (MEDI4736 - Closed to Accrual 12/2015)
Number analyzed (Participants) | 0

9. Secondary Outcome: Investigator-assessed Progression-free Survival Assessed Using a Modified Response Criteria Adapted for Immunotherapy in PD-L1 Positive Participants Treated With MEDI4736
Description: as for outcome 8
Time Frame: up to 3 years post registration
Population: No data collected for this outcome measure
Arm/Group | Arm I (MEDI4736 - Closed to Accrual 12/2015)
Number analyzed (Participants) | 0

10. Secondary Outcome: Overall Survival
Description: Duration from date of sub-study registration (or date of screening/pre-screening registration if participant never enrolls in a sub-study) to date of death due to any cause.
  Note: The docetaxel arm was closed early due to removal of docetaxel as standard of care treatment. The analyses has been restricted to participants randomized to both arms before the docetaxel arm closed.
Time Frame: Up to 3 years post registration
Population: Eligible and evaluable participants enrolled before docetaxel arm closed
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (MEDI4736 - Closed to Accrual 12/2015) | Arm II (Docetaxel - Closed to Accrual 4/2015)
Number analyzed (Participants) | 32 | 30
months | 12.1 [9.2 to 17.7] | 7.7 [6.6 to 10.7]

11. Secondary Outcome: Investigator-assessed Progression-free Survival
Description: Duration from date of sub-study registration to date of first documentation of progression, per RECIST 1.1, assessed by local review or symptomatic deterioration, or death due to any cause.
  Note: The docetaxel arm was closed early due to removal of docetaxel as standard of care treatment. The analyses has been restricted to participants randomized to both arms before the docetaxel arm closed.
Time Frame: Up to 3 years post registration
Population: Eligible and evaluable participants enrolled before docetaxel arm closed
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (MEDI4736 - Closed to Accrual 12/2015) | Arm II (Docetaxel - Closed to Accrual 4/2015)
Number analyzed (Participants) | 32 | 30
months | 3.1 [2.3 to 6.4] | 2.8 [1.4 to 4.6]

12. Secondary Outcome: Investigator-assessed Progression-free Survival Assessed Using a Modified Response Criteria Adapted for Immunotherapy
Description: Duration from date of sub-study registration to date of first documentation of progression, per RECIST 1.1, assessed by local review or symptomatic deterioration, or death due to any cause.
Time Frame: Up to 3 years post registration
Population: Data were not collected for this measure
Arm/Group | Arm I (MEDI4736 - Closed to Accrual 12/2015) | Arm II (Docetaxel - Closed to Accrual 4/2015)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Response Rate
Description: The percentage of participants with confirmed and unconfirmed, partial response and complete response to treatment with MEDI4736 or docetaxel per Response Evaluation Criteria in Solid Tumors Criteria (RECIST 1.1).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
  Note: The docetaxel arm was closed early due to removal of docetaxel as standard of care treatment. The analyses has been restricted to participants randomized to both arms before the docetaxel arm closed.
Time Frame: Up to 3 years post registration
Population: Eligible and evaluable participants enrolled before docetaxel arm closed
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (MEDI4736 - Closed to Accrual 12/2015) | Arm II (Docetaxel - Closed to Accrual 4/2015)
Number analyzed (Participants) | 32 | 30
percentage of participants | 18.8 [5.2 to 32.3] | 6.7 [0 to 15.6]

14. Other Pre Specified Outcome: Screen Success Rate
Description: Will be monitored by the percentage of screened patients that register to a therapeutic sub-study.
Time Frame: Up to 3 years
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Treatment Arm Randomization Acceptance Rate
Description: Will be monitored by the percentage of patients that receive at least one dose of the treatment they are randomized to. (Design #1)
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Description: Only 98 participants were assessed for AEs, as 9 participants on the MEDI4736 arm and 2 on the docetaxel arm were ineligible. In addition, 1 participant on the MEDI4736 arm and 6 participants on the docetaxel arm did not receive any protocol therapy, so were not evaluable for adverse events. It was pre-specified in the Study Protocol to pool the AE data from Arm I and Arm III for the purposes of Adverse Events reporting for participants who received MEDI4736.
Groups:
- Arm I & Arm III (Initial Treatment and Retreatment With MEDI4736): Arm I- Participants receive MEDI4736 (durvalumab) IV over 60 minutes on day 1. Treatment repeats every 14 days for 12 months in the absence of disease progression or unacceptable toxicity.
  Arm III-For participants assigned to Arm 1, MEDI4736: Upon evidence of progression following discontinuation of 12 months of treatment, participants may restart treatment with Arm 3, MEDI4736 for up to 12 months with the same treatment guidelines followed during the initial 12-month treatment period. Participants will only be able to restart treatment once; thus a maximum of two 12-month periods will be allowed.
  Durvalumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Arm III
  Durvalumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Arm I & Arm III (Initial Treatment and Retreatment With MEDI4736) | Arm II (Docetaxel - Closed to Accrual 4/2015)
All-Cause Mortality (participants affected / at risk) | 58/68 | 26/30
Serious Adverse Events (participants affected / at risk) | 27/68 | 3/30
Other Adverse Events (participants affected / at risk) | 66/68 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I & Arm III (Initial Treatment and Retreatment With MEDI4736) (N=68) | Arm II (Docetaxel - Closed to Accrual 4/2015) (N=30)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0
Heart failure (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1 | 0
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Infusion related reaction (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Infections and infestations-Other (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 4 | 0
Sepsis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Syncope (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I & Arm III (Initial Treatment and Retreatment With MEDI4736) (N=68) | Arm II (Docetaxel - Closed to Accrual 4/2015) (N=30)
Anemia (Blood and lymphatic system disorders) | 22 | 19
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac disorders-Other (Cardiac disorders) | 2 | 0
Chest pain - cardiac (Cardiac disorders) | 2 | 0
Heart failure (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 3 | 4
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Endocrine disorders-Other (Endocrine disorders) | 3 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 9 | 1
Hypothyroidism (Endocrine disorders) | 9 | 2
Blurred vision (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 0 | 1
Eye disorders-Other (Eye disorders) | 2 | 0
Eye pain (Eye disorders) | 1 | 0
Flashing lights (Eye disorders) | 1 | 0
Watering eyes (Eye disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Anal pain (Gastrointestinal disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 19 | 10
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 13 | 9
Dry mouth (Gastrointestinal disorders) | 6 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 4 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1 | 2
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 6
Nausea (Gastrointestinal disorders) | 22 | 11
Vomiting (Gastrointestinal disorders) | 7 | 6
Chills (General disorders) | 6 | 4
Death NOS (General disorders) | 1 | 0
Edema face (General disorders) | 2 | 1
Edema limbs (General disorders) | 10 | 5
Fatigue (General disorders) | 33 | 21
Fever (General disorders) | 7 | 3
Flu like symptoms (General disorders) | 1 | 1
Gait disturbance (General disorders) | 2 | 0
General disorders and admin site conditions - Other (General disorders) | 1 | 3
Infusion related reaction (General disorders) | 1 | 0
Injection site reaction (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 4
Non-cardiac chest pain (General disorders) | 2 | 3
Pain (General disorders) | 11 | 5
Immune system disorders-Other (Immune system disorders) | 0 | 1
Bronchial infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Infections and infestations-Other (Infections and infestations) | 5 | 1
Lung infection (Infections and infestations) | 4 | 3
Mucosal infection (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Papulopustular rash (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 2 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Fracture (Injury, poisoning and procedural complications) | 3 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 12 | 2
Alkaline phosphatase increased (Investigations) | 18 | 4
Aspartate aminotransferase increased (Investigations) | 10 | 4
Blood bilirubin increased (Investigations) | 4 | 2
Cardiac troponin I increased (Investigations) | 1 | 0
Cholesterol high (Investigations) | 1 | 0
Creatinine increased (Investigations) | 11 | 4
Ejection fraction decreased (Investigations) | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 0
INR increased (Investigations) | 3 | 0
Investigations-Other (Investigations) | 2 | 2
Lipase increased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 10 | 13
Neutrophil count decreased (Investigations) | 1 | 10
Platelet count decreased (Investigations) | 5 | 5
Serum amylase increased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 0 | 1
Weight gain (Investigations) | 3 | 1
Weight loss (Investigations) | 17 | 4
White blood cell decreased (Investigations) | 2 | 11
Alcohol intolerance (Metabolism and nutrition disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 20 | 13
Dehydration (Metabolism and nutrition disorders) | 6 | 5
Hypercalcemia (Metabolism and nutrition disorders) | 6 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 14 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 8 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 16 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 4
Hyponatremia (Metabolism and nutrition disorders) | 21 | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 | 7
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 6 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 3
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ataxia (Nervous system disorders) | 0 | 1
Concentration impairment (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 6 | 6
Dysgeusia (Nervous system disorders) | 10 | 5
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 10 | 2
Lethargy (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 2
Paresthesia (Nervous system disorders) | 2 | 1
Peripheral motor neuropathy (Nervous system disorders) | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 6
Presyncope (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 2 | 1
Tremor (Nervous system disorders) | 2 | 0
Agitation (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 4 | 1
Confusion (Psychiatric disorders) | 0 | 3
Depression (Psychiatric disorders) | 4 | 1
Insomnia (Psychiatric disorders) | 6 | 4
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 2 | 0
Hematuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 2
Renal and urinary disorders-Other (Renal and urinary disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 1
Vaginal inflammation (Reproductive system and breast disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 3
Nail loss (Skin and subcutaneous tissue disorders) | 1 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Surgical and medical procedures-Other (Surgical and medical procedures) | 1 | 0
Hot flashes (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 7 | 2
Hypotension (Vascular disorders) | 7 | 6
Phlebitis (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
Vascular disorders-Other (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT02766335/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT02766335/ICF_001.pdf